CLINICAL TRIAL: NCT03179384
Title: Impact on the Intestinal Microbiota of Treatment With Ceftriaxone in Women's Acute Community Pyelonephritis
Acronym: CEFIMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-AOI-02
Record Dates: First submitted 2017-05-29; First posted 2017-06-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pyelonephritis Acute
MeSH Terms: interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ceftriaxone treatment (Experimental)
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Ceftriaxone — ceftriaxone (1g intravenous or 1g/35mL intramuscular) will be given to patients during 7 days

SUMMARY:
Acute pyelonephritis (APN) corresponds to infections of the renal parenchyma. The annual incidence of these infections is estimated at 4-6 million cases in France, with 60 to 90% of patients managed in general city medicine. The ceftriaxone, parenteral third-generation cephalosporin (C3G), occupies an important place in the antibiotic treatment of these infections: this is the recommended probabilistic treatment, and in some situations the treatment can be continued in its entirety via a Ceftriaxone monotherapy.

The aim of the last antibiotic plan is to avoid the use of antibiotic therapies with a high selection capacity (cephalosporins, penicillins, fluoroquinolones, etc.) and thus reduce the incidence and prolongation over time of the digestive carriage of multi-resistant bacteria .

To date, there have been few studies evaluating the impact of ceftriaxone on the emergence of multi-resistant bacteria on an individual scale, with rather heterogeneous results (13-86% C3G resistance).

Thus, before considering randomized studies comparing the ecological impact of different molecules or therapeutic regimens in the treatment of ANP, it is necessary to have a precise and rigorous evaluation of the ecological impact of the molecule reference in this indication.

The investigators propose a study to evaluate the impact on the digestive flora at 1 month of a ceftriaxone antibiotic therapy (7 days) in the management of acute pyelonephritis in women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 years old
* Admitted to the emergency department with a diagnosis of PNA (simple or at risk of complications, without signs of seriousness)

Exclusion Criteria:

* Hypersensitivity to ceftriaxone, to another cephalosporin or to any of the excipients
* A history of severe hypersensitivity (eg anaphylactic reaction) to another class of antibacterial agent in the beta-lactam family (penicillins, monobatams and carbapenems)
* Severe pyelonephritis, including obstructive APN
* Pyelonephritis in patients with a urinary catheter
* Antibiotic treatment in the previous 6 months
* Chronic dialysis patient
* Patient with hepatic impairment
* Pregnancy or breast-feeding in progress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Emergence of ceftriaxone-resistant Enterobacteriaceae | at 28 days
  The emergence of ceftriaxone-resistant Enterobacteriaceae at 28 days after cessation of treatment on rectal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa DEMONCHY, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France